CLINICAL TRIAL: NCT03598842
Title: Tuberculosis- Learning the Impact of Nutrition
Brief Title: Tuberculosis - Learning the Impact of Nutrition
Acronym: TB-LION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Rutgers, The State University of New Jersey (Other); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-37473; 6005415 (Other Grant/Funding Number: Warren Alpert Foundation)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis; Malnutrition; Helminth Infection
Keywords: blood signature of Tb risk; anti Mtb immunity; RNA biomarkers; RePORT Study; India
MeSH Terms: conditions — Tuberculosis; Malnutrition; Trematode Infections | interventions — Geritol; Albendazole; Ivermectin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Malnourished without lung parasites (Experimental): Thirty study participants, household contacts of an index TB case, who are malnourished and do not have lung parasites will be consented into the study intervention. The household contact and the rest of the household members will receive nutritional supplementation meals for six months. The family will receive the food in biweekly installments and will be given a vegan meal plan.The consented household contact will also receive a daily multivitamin.
  Interventions: Dietary Supplement: Nutritional Supplementation Meal; Dietary Supplement: Multivitamin
- Malnourished with lung parasites (Experimental): Thirty study participants, household contacts of an index TB case, who are malnourished and have lung parasites will be consented into the study intervention. The household contact and the rest of the household members will receive nutritional supplementation meals for six months. The family will receive the food in biweekly installments and will be given a vegan meal plan. The consented household contact will also receive a daily multivitamin. These thirty study participants will be given anti-parasitic medications such as albendazole, ivermectin, metronidazole, or other medication per Indian guidelines to treat the parasite infection.
  Interventions: Dietary Supplement: Nutritional Supplementation Meal; Dietary Supplement: Multivitamin; Drug: Anti-parasitic medications
- Well-nourished with lung parasites (Active Comparator): These thirty study participants will be given anti-parasitic medications such as albendazole, ivermectin, metronidazole, or other medication per Indian guidelines to treat the parasite infection.
  Interventions: Drug: Anti-parasitic medications
- Well-nourished without lung parasites (No Intervention): These thirty study participants will serve as the control.These participants will be well-nourished and not have a parasite infection; therefore, they will not receive the nutritional supplementation or treatment for parasite infection.

INTERVENTIONS:
Dietary Supplement: Nutritional Supplementation Meal — Study participants will be given a nutritional supplementation for 6 months. The supplementation consists of a vegan meal plan.
  Arms: Malnourished with lung parasites; Malnourished without lung parasites
Dietary Supplement: Multivitamin — Study participants will be given a daily multivitamin to take for 6 months.
  Arms: Malnourished with lung parasites; Malnourished without lung parasites
Drug: Anti-parasitic medications — Study participants will be given anti-parasitic medications per Indian guidelines such as albendazole, ivermectin, metronidazole, or other medications to treat their parasitic infection.
  Other Names: albendazole, ivermectin, metronidazole
  Arms: Malnourished with lung parasites; Well-nourished with lung parasites

SUMMARY:
The proposed work is based on the finding that one-third of the world is infected with the bacteria Mycobacterium tuberculosis (Mtb) and only 10% of these individuals develop TB. The study aims to identify factors that drive progression to disease and study signals (markers of the immune response) that detect who will progress to active TB and why this happens. Armed with these markers, the study will address how malnutrition and worms alter this signal profile to cause active TB. The work will be conducted in India, where there are 2.8 million TB cases each year - more than any other country - and where the government has committed to eliminating TB by 2035. Data suggest that malnutrition and parasites increase risk of TB disease so the investigators will feed malnourished household contacts and have those with parasites receive medication to treat these. Using this infrastructure, the investigators will evaluate the immunologic impact of feeding on TB pathogenesis. An additional aim is to understand the role of parasitic worms with the goal of determining the utility of low-cost ($.02 per dose) worm treatment as part of TB control efforts. Risk of developing TB will be evaluated for 120 household contacts of TB patients in the setting of their malnutrition and parasites. There are four study arms comprised of thirty participants each -- malnourished with parasite infection, malnourished with no parasite infection, well-nourished with parasite infection, and well-nourished with no parasite infection. Correlates of risk of disease will be assessed using blood messenger RNA/micro RNA (mRNA/miRNA) sequencing and T cell immune markers. The TB LION study will confirm that malnutrition and worms increase the risk of active TB and will provide the basis for effective interventions that could change the face of the TB pandemic and have a profound impact on the health of people worldwide. Participants in this study will be household contacts of tuberculosis index cases. The index cases in this study do not participate in the study once a household contact is established. All interventions and follow up are only being conducted within the household contact cohort. All intervention supplies, treatments, and biologics will be purchased internationally.

ELIGIBILITY:
Inclusion Criteria: Household Contacts

* Household contact that has been housemate of eligible index case for at least the last month (See index case criteria below).
* HIV seronegative
* Willing to be tested for pregnancy if married
* Age 18-60 years
* Willingness by the patient to attend scheduled follow-up visits and undergo study assessments
* Able to provide informed consent
* Intervention inclusion: On average, one meal consumed at home per day.

Exclusion Criteria: Household Contacts

* In the team's judgement, individual is not expected to survive for 12 months
* HIV infection or not willing to undergo HIV testing (if no documented HIV test)
* Pregnant at enrollment
* Known diabetes mellitus or evidence of diabetes on hemoglobin A1C (HA1C)
* Xpert positive among those able to produce sputum
* TB symptoms (night sweats, weight loss, cough) - Only if sputum positive
* Any history of TB disease during their lifetime
* We will retrospectively exclude household contacts of presumed TB cases whose cultures do not confirm Mtb or who are Xpert negative.
* Evidence of kwashiorkor (pitting edema of foot or lower leg) those with BMI <16
* Abnormal K, Mg, Phos in those with BMI <16

Inclusion Criteria: Index Case

* Sputum Ziehl-Neelsen stain positive for acid-fast bacillus (AFB) ≥1+
* Culture or Xpert positive for Mtb; those who are smear+ but ultimately Xpert or culture negative, will be included until their culture results return at which time they will retrospectively be removed from the study.
* No history of TB treatment (i.e., no history of partial or complete treatment for a previous TB episode)
* Has at least 1 household contact with whom they have shared a house during the previous one month
* Agrees to have household contact notified about study

Exclusion Criteria: Index Case

* Pregnant at enrollment
* No Xpert or culture confirmation and unable to provide sputum sample
* No household contacts who share room
* Known Multidrug-resistant tuberculosis (MDR-TB) or extensively drug-resistant tuberculosis (XDR-TB) case
* BMI <14 kg/m2
* Abnormal K, Mg, Phos in those with BMI 14 - 16
* Lower extremity edema/kwashiorkor those with BMI 14-16
* Reported neuropathy in lower extremities (may result from thiamine deficiency)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 786 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Immune response | Visit 1
  Interferon Gamma-peripheral blood mononuclear cell (PBMC) from malnourished and well-nourished household contacts (HHC) will be labeled with carboxyfluorescein succinimidyl ester (CFSE) and then stimulated with early secreted antigen target-6 (ESAT-6) and culture filtrate protein-10 (CFP-10) peptide libraries. After 72 hours, supernatants will be harvested and the cells analyzed by flow cytometry to monitor proliferating cells. As CFSE concentrations in a cell are halved with every cell division, each generation of cells appears as a distinct peak on the flow cytometry histogram providing a proliferative index. Supernatants will be evaluated by multiplex ELISA.
Immune response | Visit 2 (approximately 7 days after visit 1)
  Interferon Gamma - PBMC from malnourished and well-nourished HHC will be labeled with carboxyfluorescein succinimidyl ester (CFSE) and then stimulated with ESAT-6 and CFP-10 peptide libraries. After 72 hours, supernatants will be harvested and the cells analyzed by flow cytometry to monitor proliferating cells. As CFSE concentrations in a cell are halved with every cell division, each generation of cells appears as a distinct peak on the flow cytometry histogram providing a proliferative index. Supernatants will be evaluated by multiplex ELISA.
Immune response | Visit 5 (3 months after parasite treatment / intervention initiation)
  Interferon Gamma - PBMC from malnourished and well-nourished HHC will be labeled with carboxyfluorescein succinimidyl ester (CFSE) and then stimulated with ESAT-6 and CFP-10 peptide libraries. After 72 hours, supernatants will be harvested and the cells analyzed by flow cytometry to monitor proliferating cells. As CFSE concentrations in a cell are halved with every cell division, each generation of cells appears as a distinct peak on the flow cytometry histogram providing a proliferative index. Supernatants will be evaluated by multiplex ELISA.
Immune Response | Visit 6 (6 months after parasite treatment / intervention initiation)
  Interferon Gamma - PBMC from malnourished and well-nourished HHC will be labeled with carboxyfluorescein succinimidyl ester (CFSE) and then stimulated with ESAT-6 and CFP-10 peptide libraries. After 72 hours, supernatants will be harvested and the cells analyzed by flow cytometry to monitor proliferating cells. As CFSE concentrations in a cell are halved with every cell division, each generation of cells appears as a distinct peak on the flow cytometry histogram providing a proliferative index. Supernatants will be evaluated by multiplex ELISA.
Immune Response | Visit 7 (12 months after parasite treatment / intervention initiation)
  Interferon Gamma - PBMC from malnourished and well-nourished HHC will be labeled with carboxyfluorescein succinimidyl ester (CFSE) and then stimulated with ESAT-6 and CFP-10 peptide libraries. After 72 hours, supernatants will be harvested and the cells analyzed by flow cytometry to monitor proliferating cells. As CFSE concentrations in a cell are halved with every cell division, each generation of cells appears as a distinct peak on the flow cytometry histogram providing a proliferative index. Supernatants will be evaluated by multiplex ELISA.

SECONDARY OUTCOMES:
Anthropometric measurement | Visit 1
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
Anthropometric measurement | Visit 5 (3 months after parasite treatment / intervention initiation)
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
Anthropometric measurement | Visit 6 (6 months after parasite treatment / intervention initiation)
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
Anthropometric measurements | Visit 7 (12 months after parasite treatment / intervention initiation)
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
Anthropometric measurements | Visit 8 (18 months after parasite treatment / intervention initiation)
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
Anthropometric measurements | Visit 9 (24 months after parasite treatment / intervention initiation)
  Body Mass Index - (BMI; weight/height in kg/m2). Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.

CONTACTS AND LOCATIONS:
Overall Officials: Pranay Sinha, MD, Principal Investigator — Boston University
Locations (1):
- Jawaharlal Institute of Postgraduate Medical Education and Research, Pondicherry, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cintron C, Narasimhan PB, Locks L, Babu S, Sinha P, Rajkumari N, Kaipilyawar V, Bhargava A, Maloomian K, Chandrasekaran P, Verma S, Joseph N, Johnson WE, Wanke C, Horsburgh CR Jr, Ellner JJ, Sarkar S, Salgame P, Lakshminarayanan S, Hochberg NS. Tuberculosis-Learning the Impact of Nutrition (TB LION): protocol for an interventional study to decrease TB risk in household contacts. BMC Infect Dis. 2021 Oct 12;21(1):1058. doi: 10.1186/s12879-021-06734-z. PMID 34641820